CLINICAL TRIAL: NCT04480476
Title: A Retrospective, Chart Review Study to Evaluate Ocular Disease Progression in Children With Late-infantile Neuronal Ceroid Lipofuscinosis Type 2 (CLN2)
Brief Title: A Retrospective, Natural History Study in Children With CLN2
Status: Withdrawn | Type: Observational
Why Stopped: study stopped due to company decision
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-381-9102
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Late-infantile Neuronal Ceroid Lipofuscinosis Type 2 (CLN2)
Keywords: CLN2, Batten Disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi center, retrospective, chart review study to document the evolution of ocular disease progression in pediatric patients with CLN2.

DETAILED DESCRIPTION:
CLN2 is a rare disease with limited available ocular natural history data. While current standard of care slows motor degeneration, it is not known to treat the ocular manifestations of disease. This study is planned to document, through retrospective data collection, ocular disease progression in children with a clinical presentation consistent with CLN2. No investigational product is administered in this retrospective, chart review study.

ELIGIBILITY:
Inclusion Criteria:

A participant is eligible to be included in the study only if all of the following criteria apply:

1. The participant's legal guardian(s) is(are) willing and able to provide them written, signed informed consent.
2. The participant has a documented diagnosis of CLN2 disease due to TPP1 deficiency, or has a relative clinically diagnosed with CLN2 disease who has the same CLN2 mutations as the participant
3. The participant has had one or more eye examinations by an eye care specialist at any time since birth.

Exclusion Criteria:

No exclusion criteria apply to this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CLN2 Batten Disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Characterize retinal structural changes in children with CLN2 | From first available medical chart through informed consent, an average of 10 years
  As assessed in by SD-OCT measures in ophthalmic records of children with CLN2

SECONDARY OUTCOMES:
Characterize changes in visual function. | From first available medical chart through informed consent, an average of 10 years
  As measured by changes in visual acuity over time in ophthalmic records of children with CLN2.

IPD SHARING:
Plan to Share IPD: No